CLINICAL TRIAL: NCT05477381
Title: Assessment of Cervical SofTening and the Prediction of Preterm Birth'
Brief Title: Cervical Softening and the Prediction of Preterm Birth
Acronym: STIPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Pregnolia AG (Industry)
Responsible Party: Principal Investigator, Martijn A. Oudijk, MD, PhD, Prof. Dr. M.A.Oudijk, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL80642.000.22
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Preterm Birth; Threatened Preterm Labor; Premature Birth; Premature Labor; Diagnosis; Cervical Incompetence, With Delivery; Cervical Incompetence in Pregnancy as Antepartum Condition
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Disease; Uterine Cervical Incompetence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic women with a history of preterm birth: Pregnant women >18 years of age, with a history of spontaneous PTB before 34 weeks. All women have biweekly visits for routine transvaginal cervical length measurement between 14-24 weeks of gestation. During these visits data on cervical softening will be collected as additional marker.
  Interventions: Diagnostic Test: Measurement of cervical stiffness by Pregnolia Device
- Symptomatic women with symptoms of threatened preterm birth: Pregnant women >18 years of age, between 24 and 34 weeks of gestation, presenting with symptoms of threatened Preterm birth (e.g. abdominal pain, blood loss, contractions, or other complaints suggestive for threatened Preterm birth).
  Interventions: Diagnostic Test: Measurement of cervical stiffness by Pregnolia Device

INTERVENTIONS:
Diagnostic Test: Measurement of cervical stiffness by Pregnolia Device — The Pregnolia® System is designed to provide information about the mechanical properties of the cervical tissue by assessing the CSI (Cervical Stiffness Index) through a probe that will create a weak vacuum to retract tissue. The Pregnolia® System is designed with the purpose to provide an alternative diagnostic marker to identify women at risk of spontaneous PTB.
  The Pregnolia® System is a CE-marked device developed for quantitative assessment of softening of the uterine cervix.
  The Pregnolia® System will be applied within its intended use.

SUMMARY:
Currently, transvaginal cervical length measurement is used to screen in asymptomatic pregnant women with a history of PTB. In symptomatic women, presenting with threatened PTB cervical length in combination with the fibronectin test is used to identify women at high risk to deliver preterm. However, the predictive capacity of transvaginal cervical length measurement is limited. In pregnant women with a history of PTB, it only identifies a proportion of women who will have recurrent PTB. For symptomatic women, 30-60% of these women admitted to the hospital, do not deliver within seven days, leading to overtreatment of these women.

Cervical softening is precursor of cervical shortening, effacement and dilatation and therefore cervical softening is a promising new marker that is based on tissue elasticity. However, the predictive value of cervical softening and the relation with spontaneous PTB still has to be determined. With the newly developed Pregnolia® System cervical softness could be measured on a standardized and safe manner. This study could help to improve care for women with a history of spontaneous PTB.

DETAILED DESCRIPTION:
Preterm birth (PTB) is amongst the leading causes of perinatal and childhood morbidity and mortality. Therefore, accurate identification of pregnant women at high risk of PTB is important. Identifying these women, enables obstetric healthcare professionals to apply interventions to postpone delivery and/or to prevent PTB to improve perinatal and childhood outcomes.

Currently, transvaginal cervical length measurement is used to screen asymptomatic pregnant women with a history of PTB to identify women requiring a cerclage. In symptomatic women, presenting with threatened (PTB), cervical length in combination with the fetal fibronectin(fFN) test is used to identify women at high risk to deliver within 7 days of presentation. However, the predictive capacity of transvaginal cervical length measurement is limited. In pregnant women with a history of PTB, it only identifies a proportion of women who will have recurrent PTB. For symptomatic women, 30-60% of these women admitted to the hospital, do not deliver within seven days, leading to overtreatment of these women.

Since cervical softening is a precursor of cervical shortening, effacement and dilatation, cervical softening is a promising new marker that is based on tissue elasticity. It can be measured with the CE-marked Pregnolia® System for accurate characterization of cervical softening status. It provides a value for tissue elasticity on a continuous scale.

A previous study has shown that softening of the cervix can be detected before shortening of the cervix. The Pregnolia® System may allow to detect women at risk for PTB earlier compared to traditional transvaginal ultrasound that measures shortening of the cervix, and therefore may prove useful for a more accurate risk assessment of PTB.

This current study is a single centre cohort study, where Two cohorts of women will be investigated. 1) Asymptomatic pregnant women with a history of spontaneous PTB before 34 weeks of gestation (Cohort A-STIPP). 2) Symptomatic women presenting with threatened PTB between 24 and 34 weeks (Cohort S-STIPP).

Objective: The aim of this study is to evaluate the predictive capacity of cervical softening and risk of PTB.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above.
* Ability to understand Dutch or English (both spoken and written).
* Ultrasound-based gestational age determined by measurement of crown rump length (CRL) determined between 9 and 11 weeks of gestation.
* Singleton and twin pregnancies.

Cohort A-STIPP specific:

- Medical history of spontaneous preterm birth before 34 weeks of gestation

Cohort S-STIPP specific:

* Threatened Preterm birth between 24 and 34 weeks of gestation.
* Threatened preterm birth is defined as:

  * abdominal pain
  * (Braxton Hicks) contractions
  * vaginal blood loss.

Exclusion Criteria:

* Under 18 years of age.
* Signs of intrauterine infection.
* Obstetric indication for immediate delivery (advanced labor, cord prolapse, abruption, signs of fetal distress).
* Confirmed fetal abnormality.
* Confirmed preterm rupture of membranes.
* Confirmed vasa / placenta praevia.
* Severe vaginal bleeding and light bleeding that cannot be stopped.
* Signs of imminent labor such as blood loss, regular contractions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes pregnant women
Study Population: Women with an increased risk of preterm birth. Women are eligible when they fall in one of following categories:
  * Medical History of Spontaneous Preterm Birth before 34 weeks of gestation or
  * Threatened Preterm Birth between 24 and 34 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Preterm Birth < 34 weeks | Maximum time frame up to 28 weeks: from inclusion at 14 weeks of gestational age until delivery, with a maximum of 42 weeks of gestational age.
  Spontaneous preterm birth before 34 weeks of gestation in the asymptomatic cohort
Delivery within seven days after inclusion | From inclusion until 7 days later
  Delivery within seven days after inclusion in the symptomatic cohort

SECONDARY OUTCOMES:
Spontaneous preterm birth <37 weeks | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Spontaneous preterm birth <37 weeks of gestational age
Spontaneous preterm birth <34 weeks | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Spontaneous preterm birth <34 weeks of gestational age
Spontaneous preterm birth <32 weeks | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Spontaneous preterm birth <32 weeks of gestational age
Spontaneous preterm birth <28 weeks | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Spontaneous preterm birth <28 weeks of gestational age
Prediction of preterm birth using cervical softening. | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Development of a prediction model using cervical softening to predict the risk of preterm birth before 37, 34, 32 and 28 weeks.
Prediction of preterm birth using the combination of cervical softening and transvaginal cervical length measurement. | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Development of a prediction model using the combination of cervical softening and transvaginal cervical length measurement to predict the risk of preterm birth before 37, 34, 32 and 28 weeks.
Prediction of preterm birth using the combination of cervical softening, transvaginal cervical length measurement, and fetal fibronectin. | From inclusion (symptomatic cohort 24-34 weeks) until delivery with a maximum of 42 weeks of gestational age
  Development of a prediction model using the combination of cervical softening, transvaginal cervical length measurement, and fetal fibronectin to predict the risk of preterm birth before 37, 34, 32 and 28 weeks. (only for symptomatic women)
Prediction of latency time using cervical softening. | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age
  Development of a prediction model using cervical softening to predict the latency time (interval between inclusion and delivery).
Prediction of latency time using the combination of cervical softening and transvaginal cervical length measurement. | From inclusion (symptomatic cohort 24-34 weeks, asymptomatic cohort 14 weeks) until delivery with a maximum of 42 weeks of gestational age.
  Development of a prediction model using the combination of cervical softening and transvaginal cervical length measurement to predict the latency time (interval between inclusion and delivery).
Prediction of latency time using the combination of cervical softening, transvaginal cervical length measurement, and fetal fibronectin | From inclusion (symptomatic cohort 24-34 weeks) until delivery with a maximum of 42 weeks of gestational age.
  Development of a prediction model using the combination of cervical softening, transvaginal cervical length measurement, and fetal fibronectin to predict the latency time. (interval between inclusion and delivery). (only for symptomatic women)

OTHER OUTCOMES:
Patient discomfort of Pregnolia measurement | In asymptomatic cohort at 14, 16, 18, 20, 22 and 24 weeks of gestational age, in the symptomatic cohort at moment of inclusion
  Pain during Pregnolia measured on a visual analogue scale (VAS) from "no pain"to "worst possible pain"
Vaginal or Cervical blood loss (directly after measurement) | In asymptomatic cohort at 14, 16, 18, 20, 22 and 24 weeks of gestational age, in the symptomatic cohort at moment of inclusion
  Vaginal or Cervical blood loss, noticed directly (= within 30 minutes) after measurement
Infections within seven days of measurement | From inclusion up to 1 week
  Infections within seven days of measurement (urinary tract infections, vaginal infections, intra-uterine infections)
Preterm Prelabour Rupture of membranes at moment of measurement | Within 1 hour after measurement
  Preterm Prelabour Rupture of membranes at moment of measurement
Irritation and sensitization of mucosal tissue | Within 1 hour after measurement
  Irritation and sensitization of mucosal tissue as noticed by the researcher performing the measurement
Superficial lacerations or minor tissue abrasions | Within 1 hour after measurement
  Superficial lacerations or minor tissue abrasions

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pajkrt, Prof. Dr., Principal Investigator — Amsterdam UMC, location AMC; Martijn Oudijk, Prof. Dr., Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All agreements regarding data sharing are defined in a signed Clinical Trial Agreement (CTA), GDPR are applicable to this agreement.
Supporting Information: Study Protocol, CSR
Time Frame: After publication of the manuscript
Access Criteria: Data are available upon reasonable request

REFERENCES:
- [Derived] Breuking S, Oudijk MA, van Eekelen R, de Boer MA, Pajkrt E, Hermans F. Assessment of cervical softening and the prediction of preterm birth (STIPP): protocol for a prospective cohort study. BMJ Open. 2023 Nov 21;13(11):e071597. doi: 10.1136/bmjopen-2023-071597. PMID 37989370